CLINICAL TRIAL: NCT03629340
Title: Phase II Trial of Metformin for Pulmonary Hypertension in Heart Failure With Preserved Ejection Fraction
Brief Title: Metformin for Pulmonary Hypertension HFpEF
Acronym: PH-HFpEF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY19020231; R01AG058659 (NIH)
Record Dates: First submitted 2018-08-10; First posted 2018-08-14 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Pulmonary Hypertension; Heart Failure
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Drug: Metformin (Experimental): 500mg PO (by mouth) BID (two times daily) x 1 week then increase to 1000mg PO BID x 11 weeks
  Interventions: Drug: Metformin
- Placebo Oral Capsule (Placebo Comparator): Placebo capsule that is of identical size, shape, and color to experimental drug capsule PO (by mouth) BID (two times each day) for 12 weeks
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Metformin — 500 mg PO BID x 1 week then increase to 1000 mg PO BID x 11 weeks
  Arms: Drug: Metformin
Drug: Placebo oral capsule — Placebo capsule that is of identical size, shape, and color to experimental drug capsule PO (by mouth) BID (two times each day) for 12 weeks
  Arms: Placebo Oral Capsule

SUMMARY:
The main objective of this study is to determine the clinical efficacy of metformin versus placebo and the therapeutic response with regards to functional capacity and hemodynamics in PH-HFpEF.

DETAILED DESCRIPTION:
This is a 12-week blinded cross over trial of metformin in PH-HFpEF to improve exercise hemodynamics, functional capacity, and glucose metabolism. This phase II clinical trial will provide detailed phenotyping, physiological and mechanistic data on PH-HFpEF.

ELIGIBILITY:
Inclusion Criteria:

2. PH-HFpEF Confirmed diagnosis by RHC within the past 6 months:

Mean Pulmonary Arterial Pressure (mPAP) ≥ 25 mm Hg AND Pulmonary artery wedge pressure (PAWP) ≥ 15 mm Hg AND Transpulmonary Gradient (TPG) ≥ 12 mm Hg

OR Exercise measurements

Mean Pulmonary Arterial Pressure (mPAP) ≥ 30 mm Hg AND Pulmonary artery wedge pressure (PAWP) ≥ 20 mm Hg AND PA calculation (change in mPAP/change in cardiac output) = ≥3 mmHg/L/min

3. Three or more features of metabolic syndrome defined as:

Body Mass Index (BMI) ≥ 30 kg/m² Systolic blood pressure (BP) ≥ 130 mm Hg and/or diastolic BP ≥ 85 mm Hg Elevated waist circumference > 102 cm in men and > 88 cm in women Fasting triglyceride (TG) level over 150 mg/dl High-density lipoprotein <40 mg/dL in men or < 50 mg/dL in women

Exclusion Criteria:

1. Age less than 18 years;
2. Uncontrolled systemic hypertension based on repeated measurement of sitting systolic blood pressure >170 mm Hg or sitting diastolic blood pressure >95 mm Hg at Screening;
3. Systemic sitting blood pressure < 110 mmHg systolic or < 60 mm Hg diastolic at Screening;
4. Hemoglobin A1C > 10;
5. Currently taking metformin or history of intolerance to metformin or contraindication to taking metformin;
6. Known type 1 diabetes
7. Positive urine pregnancy test or breastfeeding
8. Ejection Fraction < 50%
9. Dementia;

11. End-stage malignancy; 12. Major cardiovascular event or procedure within 6 weeks prior to enrollment; 13. Severe valvular disease; 14. Other severe acute or chronic medical, psychiatric or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study or would prevent completion of the study; 15. Current Smoker; 16. Hemoglobin <9 g/dL; 17. Estimated glomerular filtration rate (eGFR) <30 mL/min/1.73 m2; 18. Receipt of an investigational product or device, or participation in a drug research study within a period of 15 days 19. <3 months of stable dose of PDE5i

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-02-26 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the trial will be mean pulmonary artery pressure (mPAP) during submaximal exercise as compared between placebo and metformin at 12 weeks (i.e. the week 12 RHC of placebo vs week 12 RHC of metformin). | 12 weeks (i.e. the 12th week of placebo vs 12th week of metformin)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Risbano, MD, MA, Principal Investigator — University of Pittsburgh; Marc A Simon, MD, MS, Study Director — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Medical Center, San Francisco, California
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No